CLINICAL TRIAL: NCT01173263
Title: Effect of BIS Titrated Propofol Sedation on Lower Esophageal Sphincter Pressures and Esophageal Function in Intensive Care Patients
Brief Title: Effect of Bispectral Index (BIS) Titrated Propofol Sedation on Lower Esophageal Sphincter Pressures and Esophageal Function in Intensive Care Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Alparslan Turan, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-226
Record Dates: First submitted 2010-07-21; First posted 2010-08-02 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Respiration, Artificial
Keywords: breathing machine; mechanical ventilator
MeSH Terms: conditions — Respiratory Aspiration | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BIS 70 (Active Comparator): BIS levels of 70, will be targeted (Anxiolysis/high-frequency EEG activity, beta-augmentation);
  Interventions: Other: BIS 70 maintained
- BIS 50 (Active Comparator): BIS levels of 50 will be targeted, (Low frequency EEG activity, theta-delta activity)
  Interventions: Other: BIS level 50
- BIS 35 (Active Comparator): BIS levels of 35 will be targeted (low frequency EEG activity)
  Interventions: Other: BIS 35

INTERVENTIONS:
Other: BIS 70 maintained — Each patient will receive propofol sedation by continuous infusion titrated to a BIS level of 70.
  Other Names: sedation; propofol; BIS monitor; esophageal pressure; esophageal function
  Arms: BIS 70
Other: BIS level 50 — Each patient will receive propofol sedation by continuous infusion titrated to a BIS level of 50.
  Other Names: sedation; propofol; BIS monitor; esophageal pressure; esophageal function
  Arms: BIS 50
Other: BIS 35 — Each patient will receive propofol sedation by continuous infusion titrated to a BIS level of 35.
  Other Names: sedation; propofol; BIS monitor; esophageal pressure; esophageal function
  Arms: BIS 35

SUMMARY:
Eligible patients will be allocated to receive propofol sedation titrated to 3 different Bispectral Index (BIS) levels in a random order. Primary hypothesis: Deepening propofol sedation - as determined by BIS - lowers esophageal pressure in critical care patients.

DETAILED DESCRIPTION:
Patient will be selected from the ICU, based on the defined inclusion and exclusion criteria. Potential study subjects will be screened by the research fellow or the on-site study co-investigator. Eligible patients will be allocated to receive propofol sedation titrated to 3 different BIS levels in a random order. BIS XP monitors (Aspect Medical Systems, Norwood, MA, USA) will be used which are relatively resistant to EMG artifact; a BIS sensor will be position on forehead of the patient after the skin is degreased and gently abraded. Esophageal pressure monitoring will be performed by a catheter inserted from the nose to the esophagus and left there trough the study period.

If patients are on sedation they will be placed on propofol sedation for a washout period. Each patient will receive propofol sedation by continuous infusion titrated to a different levels of BIS in a randomized fashion according to a computer-generated random-number sequence;

1. BIS levels of 70, will be targeted (Anxiolysis/high-frequency EEG activity, beta-augmentation);
2. BIS levels of 50 will be targeted, (Low frequency EEG activity, theta-delta activity);
3. BIS levels of 35 will be targeted (low frequency EEG activity). A propofol infusion will be titrated by the investigators to the designated BIS target according to randomization. Clinical personnel will not be blinded to the study, and if patient has clinically significant change in hemodynamic parameters study will be interrupted. Each BIS target level will be kept as constant as possible for at least one hour; thereafter, lower esophageal pressures will be recorded for 15 minutes using high resolution esophageal manometry. Studies will be done in supine position [Most ICU patients are now kept head-up.], and the manometric assembly will be positioned to record from the hypopharynx to the stomach with 4-6 of the sensors positioned in the stomach.

All patients will otherwise receive routine ICU care and medications without interruption of standard clinical care.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Written informed consent from relatives
* Clinically stable
* Mechanically ventilated < 2days
* Require sedation and expected to be given propofol

Exclusion Criteria:

* Recent injury or other pathologic condition of the esophagus
* Major bronchopleural fistula
* History of liver failure
* History of renal failure
* History of major neuromuscular disease
* Multiple trauma
* Upper motor nerve injury
* Hypersensitivity to propofol
* Recent gastrointestinal surgery
* Patients with a diagnosed or suspected condition that may give false results in BIS monitoring.
* Tracheostomized patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Deepening propofol sedation - as determined by BIS - lowers esophageal pressure in critical care patients. | for 15 minutes after assigned BIS level has been maintained for one hour, while in the ICU
  Sedation will also be evaluated with the bispectral index of the electroencephalogram. BIS of the EEG data will be acquired with 4 BIS-sensor electrodes and a BIS XP monitor. The BIS will be recorded electronically at one-minute intervals. Heart rate, blood pressures (diastolic and systolic), respiratory rate, core temperature and oxygen saturation will be recorded every 5 minutes during the measurement period of the study.

SECONDARY OUTCOMES:
Deepening propofol sedation - as measured by Sedation Agitation Scale, Richmond Agitation Scale Score, and Ramsay sedation scale - lowers esophageal pressure in critical care patients. | every 10 minutes, while sedated in the ICU
  The SAS uses a 1 to 7 point scale to make a determination of the patient's level of agitation and sedation from a rating of 7 dangerously agitated to a rating of 1 unarousable (Table 1). Clinical sedation assessments using SAS and RASS scales will be measured every 10 minutes through the study period.
Modifying the target level of BIS titration affects upper esophageal pressures and esophageal peristalsis. | for 15 minutes after assigned BIS level has been maintained for one hour, while in the ICU
  Upper esophageal sphincter pressures, transient LES relaxations, and regurgitations will be evaluated by the GI team from recorded data from high resolution manometry.
There is an association between ventilator associated pneumonia and baseline lower esophageal and barrier pressure. | daily, until hospital discharge
  Patients will be followed for their stay in the hospital for occurrence of ventilator associated pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States